CLINICAL TRIAL: NCT00439777
Title: Oral Direct Factor Xa Inhibitor Rivaroxaban in Patients With Acute Symptomatic Deep-Vein Thrombosis or Pulmonary Embolism
Brief Title: Oral Direct Factor Xa Inhibitor Rivaroxaban in Patients With Acute Symptomatic Pulmonary Embolism - The EINSTEIN PE Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Collaborators: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11702b; 2006-004495-13 (EudraCT Number)
Record Dates: First submitted 2007-02-23; First posted 2007-02-26 (Estimated); Results first posted 2013-01-24 (Estimated); Last update posted 2014-02-27 (Estimated); Status verified 2014-01

CONDITIONS: Pulmonary Embolism
MeSH Terms: conditions — Pulmonary Embolism | interventions — Rivaroxaban

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Rivaroxaban (Xarelto, BAY59-7939) (Experimental): Participants received 15 mg rivaroxaban (oral) twice daily (b.i.d.) for 3 weeks, followed by 20 mg once daily (o.d.)
  Interventions: Drug: Rivaroxaban (Xarelto, BAY59-7939)
- Enoxaparin/VKA (Active Comparator): Participants received enoxaparin (subcutaneous) 1.0 mg/kg b.i.d. for minimal 5 days, plus vitamin K antagonist (VKA) at individually titrated doses to achieve a target international normalized ratio (INR) of 2.5 (range: 2.0 - 3.0)
  Interventions: Drug: Enoxaparin overlapping with and followed by VKA

INTERVENTIONS:
Drug: Rivaroxaban (Xarelto, BAY59-7939) — During the first 3 weeks patients will receive 15 mg rivaroxaban twice-daily. Thereafter, patients will receive rivaroxaban 20 mg once-daily. Rivaroxaban will be administered orally and should be taken with food.
  Arms: Rivaroxaban (Xarelto, BAY59-7939)
Drug: Enoxaparin overlapping with and followed by VKA — Enoxaparin 1.0 mg/kg twice daily with a minimal duration of 5 days. This 5 days treatment could include the period up to 36 hr before randomization if enoxaparin twice-daily was used. VKA should be started as soon as possible but not later than 48 hours after randomization.
  Arms: Enoxaparin/VKA

SUMMARY:
This is a multicenter, randomized, open-label, assessor-blind, event-driven, non-inferiority program for efficacy with a study treatment duration of 3, 6 or 12 months in patients with confirmed acute symptomatic pulmonary embolism (PE) with or without symptomatic Deep-Vein Thrombosis (DVT) (Einstein-PE).

DETAILED DESCRIPTION:
Within the US 'Johnson & Johnson Pharmaceutical Research & Development, L.L.C.' is sponsor.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed acute symptomatic proximal PE with or without symptomatic DVT

Exclusion Criteria:

* Legal lower age limitations (country specific)
* Thrombectomy, insertion of a caval filter, or use of a fibrinolytic agent to treat the current episode of DVT and/or PE
* Other indication for VKA than DVT and/or PE
* The pre-randomization anti-coagulant treatment (Criteria # 4) has been prolonged from 36 hours to a maximum of 48 hours.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4833 (Actual)
Dates: Start 2007-03; Primary Completion 2011-09 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (254):
- United States (21):
  - Little Rock, Arkansas
  - Redlands, California
  - Bay Pines, Florida
  - Miami, Florida
  - Idaho Falls, Idaho
  - Covington, Louisiana
  - Baltimore, Maryland
  - Boston, Massachusetts
  - Chesterfield, Missouri
  - Albuquerque, New Mexico
  - Chapel Hill, North Carolina
  - Greensboro, North Carolina
  - Oklahoma City, Oklahoma
  - Camp Hill, Pennsylvania
  - Pittsburgh, Pennsylvania
  - San Antonio, Texas
  - Murray, Utah
  - Salt Lake City, Utah
  - Fredericksburg, Virginia
  - Spokane, Washington
  - Tacoma, Washington
- Les Escaldes, Andorra
- Australia (19):
  - Garran, Australian Capital Territory
  - Gosford, New South Wales
  - Kogarah, New South Wales
  - Lismore, New South Wales
  - St Leonards, New South Wales
  - Sydney, New South Wales
  - Brisbane, Queensland
  - Redcliffe, Queensland
  - Southport, Queensland
  - Woolloongabba, Queensland
  - Adelaide, South Australia
  - Woodville South, South Australia
  - Launceston, Tasmania
  - Box Hill, Victoria
  - Clayton, Victoria
  - Geelong, Victoria
  - Melbourne, Victoria
  - Fremantle, Western Australia
  - Perth, Western Australia
- Austria (5):
  - Graz, Styria
  - Vienna, Vienna
  - Feldkirch, Vorarlberg
  - Innsbruck
  - Linz
- Belgium (12):
  - Aalst
  - Bruxelles - Brussel
  - Duffel
  - Genk
  - Ghent
  - Hasselt
  - Leuven
  - Lier
  - Liège
  - Namur
  - Yvoir
  - Zottegem
- Brazil (6):
  - Curitiba, Paraná
  - Londrina, Paraná
  - Botucatu, São Paulo
  - São Paulo, São Paulo
  - Sorocaba, São Paulo
  - Rio de Janeiro
- Canada (4):
  - Winnipeg, Manitoba
  - London, Ontario
  - Ottawa, Ontario
  - Toronto, Ontario
- China (9):
  - Guangzhou, Guangdong
  - Nanning, Guangxi
  - Harbin, Heilongjiang
  - Wuhan, Hubei
  - Suzhou, Jiangsu
  - Shenyang, Liaoning
  - Hangzhou, Zhejiang
  - Beijing
  - Shanghai
- Czechia (6):
  - Kladno
  - Ostrava
  - Ostrava-Poruba
  - Prague
  - Rakovník
  - Usti Nad Lebem
- Denmark (3):
  - Aarhus C
  - Brædstrup
  - Frederiksberg
- Tallinn, Estonia
- Finland (2):
  - Tampere
  - Turku
- France (30):
  - Agen
  - Amiens
  - Angers
  - Arras
  - Besançon
  - Bordeaux
  - Brest
  - Castelnau-le-Lez
  - Clamart
  - Clermont-Ferrand
  - Colombes
  - Dijon
  - Grenoble
  - Limoges
  - Metz-Tessy
  - Montpellier
  - Nantes
  - Nice
  - Orthez
  - Paris
  - Pierre-Bénite
  - Roanne
  - Rouen
  - Saint-Etienne
  - Strasbourg
  - Toulon
  - Toulouse
  - Valenciennes
  - Vandœuvre-lès-Nancy
  - Vernon
- Germany (23):
  - Bruchsal, Baden-Wurttemberg
  - Heidelberg, Baden-Wurttemberg
  - Karlsbad, Baden-Wurttemberg
  - Neckargemünd, Baden-Wurttemberg
  - Tübingen, Baden-Wurttemberg
  - Augsburg, Bavaria
  - München, Bavaria
  - Würzburg, Bavaria
  - Hamburg, Hamburg
  - Darmstadt, Hesse
  - Frankfurt am Main, Hesse
  - Rotenburg (Wümme), Lower Saxony
  - Greifswald, Mecklenburg-Vorpommern
  - Essen, North Rhine-Westphalia
  - Paderborn, North Rhine-Westphalia
  - Witten, North Rhine-Westphalia
  - Mainz, Rhineland-Palatinate
  - Dresden, Saxony
  - Halle, Saxony-Anhalt
  - Magdeburg, Saxony-Anhalt
  - Berlin, State of Berlin
  - Nordhausen, Thuringia
  - Bottrop
- Hong Kong (2):
  - Hong Kong
  - Wan Chai
- Hungary (9):
  - Budapest
  - Debrecen
  - Kecskemét
  - Kistarcsa
  - Miskolc
  - Szekszárd
  - Szentes
  - Szombathely
  - Zalaegerszeg
- India (4):
  - Kochi, Kerala
  - Hyderabad
  - New Delhi
  - Pune
- Indonesia (5):
  - Jakarta, Indonesia
  - Bandung
  - Jakarta
  - Medan
  - Semarang
- Ballinasloe, Co. Galway, Ireland
- Israel (11):
  - Haifa, Israel
  - Holon, Israel
  - Jerusalem, Israel
  - Petah Tikva, Israel
  - Afula
  - Ashkelon
  - Haifa
  - Kfar Saba
  - Rehovot
  - Safed
  - Tel Aviv
- Italy (12):
  - Rozzano, Milano
  - Bologna
  - Chieti
  - Milan
  - Padua
  - Palermo
  - Parma
  - Pavia
  - Piacenza
  - Reggio Emilia
  - Varese
  - Venezia
- Liepāja, Latvia
- Lithuania (2):
  - Kaunas
  - Vilnius
- Kuala Selangor, Malaysia
- Netherlands (7):
  - Amsterdam
  - Arnhem
  - Enschede
  - Groningen
  - Hoofddorp
  - Maastricht
  - Zwolle
- New Zealand (4):
  - Auckland
  - Christchurch
  - Palmerston North
  - Wellington South
- Norway (4):
  - Fredrikstad
  - Oslo
  - Rud
  - Trondheim
- Quezon City, Philippines
- Poland (8):
  - Bialystok
  - Krakow
  - Lodz
  - Lublin
  - Poznan
  - Torun
  - Warsaw
  - Wroclaw
- San Juan, Puerto Rico
- Singapore, Singapore
- South Africa (6):
  - Johannesburg, Gauteng
  - Pretoria, Gauteng
  - Roodepoort, Gauteng
  - Cape Town, Western Cape
  - Somerset West, Western Cape
  - Worcester, Western Cape
- South Korea (4):
  - Seoul, Korea
  - Daegu
  - Seoul
  - Taegu
- Spain (8):
  - Barcelona, Barcelona
  - Terrassa, Barcelona
  - Valladolid, Castille and León
  - Girona, Girona
  - Palma de Mallorca, Illes Baleares
  - Madrid, Madrid
  - Pamplona, Pamplona
  - Requena, Valencia
- Sweden (5):
  - Borås
  - Gothenburg
  - Jönköping
  - Stockholm
  - Sundsvall
- Switzerland (6):
  - Bern, Canton of Bern
  - Lausanne, Canton of Vaud
  - Zurich, Canton of Zurich
  - Genéve 14, Genève 14
  - Chur, Kanton Graubünden
  - Lucerne
- Taiwan (2):
  - Taichung
  - Taipei
- Thailand (3):
  - Pathumwan, Bangkok, Thailand
  - Bangkok
  - Chiang Mai
- United Kingdom (4):
  - Plymouth, Devon
  - Isleworth, London
  - London, London
  - London

REFERENCES:
- [Result] EINSTEIN-PE Investigators; Buller HR, Prins MH, Lensin AW, Decousus H, Jacobson BF, Minar E, Chlumsky J, Verhamme P, Wells P, Agnelli G, Cohen A, Berkowitz SD, Bounameaux H, Davidson BL, Misselwitz F, Gallus AS, Raskob GE, Schellong S, Segers A. Oral rivaroxaban for the treatment of symptomatic pulmonary embolism. N Engl J Med. 2012 Apr 5;366(14):1287-97. doi: 10.1056/NEJMoa1113572. Epub 2012 Mar 26. PMID 22449293
- [Result] Prins MH, Lensing AW. Derivation of the non-inferiority margin for the evaluation of direct oral anticoagulants in the treatment of venous thromboembolism. Thromb J. 2013 Jul 6;11(1):13. doi: 10.1186/1477-9560-11-13. PMID 23829521
- [Result] Prins MH, Lensing AW, Bauersachs R, van Bellen B, Bounameaux H, Brighton TA, Cohen AT, Davidson BL, Decousus H, Raskob GE, Berkowitz SD, Wells PS; EINSTEIN Investigators. Oral rivaroxaban versus standard therapy for the treatment of symptomatic venous thromboembolism: a pooled analysis of the EINSTEIN-DVT and PE randomized studies. Thromb J. 2013 Sep 20;11(1):21. doi: 10.1186/1477-9560-11-21. PMID 24053656
- [Result] Wang Y, Wang C, Chen Z, Zhang J, Liu Z, Jin B, Ying K, Liu C, Shao Y, Jing Z, Meng IL, Prins MH, Pap AF, Muller K, Lensing AW; Chinese EINSTEIN Investigators. Rivaroxaban for the treatment of symptomatic deep-vein thrombosis and pulmonary embolism in Chinese patients: a subgroup analysis of the EINSTEIN DVT and PE studies. Thromb J. 2013 Dec 16;11(1):25. doi: 10.1186/1477-9560-11-25. PMID 24341332
- [Result] van Bellen B, Bamber L, Correa de Carvalho F, Prins M, Wang M, Lensing AW. Reduction in the length of stay with rivaroxaban as a single-drug regimen for the treatment of deep vein thrombosis and pulmonary embolism. Curr Med Res Opin. 2014 May;30(5):829-37. doi: 10.1185/03007995.2013.879439. Epub 2014 Jan 22. PMID 24432872
- [Derived] Dobesh PP, Volkl AA, Pap AF, Damaraju CV, Levitan B, Yuan Z, Amin AN. Benefit-Risk Assessment of Rivaroxaban in Older Patients With Nonvalvular Atrial Fibrillation or Venous Thromboembolism. Drugs Aging. 2025 May;42(5):469-484. doi: 10.1007/s40266-025-01192-7. Epub 2025 Mar 31. PMID 40163217
- [Derived] Ten Cate H, Lensing AWA, Weitz JI, Middeldorp S, Beyer-Westendorf J, Kubitza D, Brighton T, Raskob GE, Mismetti P, Prandoni P, Gebel M, Prins MH. The prothrombin time does not predict the risk of recurrent venous thromboembolism or major bleeding in rivaroxaban-treated patients. Thromb Res. 2018 Oct;170:75-83. doi: 10.1016/j.thromres.2018.08.008. Epub 2018 Aug 15. PMID 30121419
- [Derived] Di Nisio M, Vedovati MC, Riera-Mestre A, Prins MH, Mueller K, Cohen AT, Wells PS, Beyer-Westendorf J, Prandoni P, Bounameaux H, Kubitza D, Schneider J, Pisters R, Fedacko J, Fontes-Carvalho R, Lensing AW. Treatment of venous thromboembolism with rivaroxaban in relation to body weight. A sub-analysis of the EINSTEIN DVT/PE studies. Thromb Haemost. 2016 Sep 27;116(4):739-46. doi: 10.1160/TH16-02-0087. Epub 2016 Aug 18. PMID 27535349
- [Derived] Prins MH, Lensing AW, Brighton TA, Lyons RM, Rehm J, Trajanovic M, Davidson BL, Beyer-Westendorf J, Pap AF, Berkowitz SD, Cohen AT, Kovacs MJ, Wells PS, Prandoni P. Oral rivaroxaban versus enoxaparin with vitamin K antagonist for the treatment of symptomatic venous thromboembolism in patients with cancer (EINSTEIN-DVT and EINSTEIN-PE): a pooled subgroup analysis of two randomised controlled trials. Lancet Haematol. 2014 Oct;1(1):e37-46. doi: 10.1016/S2352-3026(14)70018-3. Epub 2014 Sep 28. PMID 27030066
- [Derived] Bauersachs RM, Lensing AW, Prins MH, Kubitza D, Pap AF, Decousus H, Beyer-Westendorf J, Prandoni P. Rivaroxaban versus enoxaparin/vitamin K antagonist therapy in patients with venous thromboembolism and renal impairment. Thromb J. 2014 Nov 24;12:25. doi: 10.1186/1477-9560-12-25. eCollection 2014. PMID 25750589
- [Derived] Wells PS, Gebel M, Prins MH, Davidson BL, Lensing AW. Influence of statin use on the incidence of recurrent venous thromboembolism and major bleeding in patients receiving rivaroxaban or standard anticoagulant therapy. Thromb J. 2014 Nov 26;12:26. doi: 10.1186/1477-9560-12-26. eCollection 2014. PMID 25698905
- [Derived] Cohen AT, Dobromirski M. The use of rivaroxaban for short- and long-term treatment of venous thromboembolism. Thromb Haemost. 2012 Jun;107(6):1035-43. doi: 10.1160/TH11-12-0859. Epub 2012 Feb 28. PMID 22371186

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with confirmed acute symptomatic pulmonary embolism (PE) with or without symptomatic deep vein thrombosis (DVT) were recruited at specialized study sites.
Pre-assignment Details: Out of 4843 participants screened, 10 failed screening (6 due to protocol violations, 2 due to investigator decision and another 2 subjects due to technical problems [interactive voice response system did not work properly]). 4833 participants were randomized (2420 to rivaroxaban and 2413 to enoxaparin/VKA).
Period: Treatment Period
Arm/Group | Rivaroxaban (Xarelto, BAY59-7939) | Enoxaparin/VKA
Started | 2420 | 2413
Participants Received Treatment | 2412 | 2405
Completed | 2001 | 1954
Not Completed | 419 | 459
Not completed — Death | 29 | 21
Not completed — Study terminated by sponsor | 125 | 132
Not completed — Site closed by investigator | 0 | 1
Not completed — Did not take study treatment | 7 | 8
Not completed — Adverse Event | 111 | 92
Not completed — Protocol Violation | 23 | 30
Not completed — Withdrawal by Subject | 66 | 118
Not completed — Lack of Efficacy | 1 | 4
Not completed — Lost to Follow-up | 8 | 10
Not completed — Protocol driven decision point | 1 | 3
Not completed — Physician Decision | 7 | 18
Not completed — Clinical endpoint reached | 26 | 13
Not completed — Technical problems | 3 | 1
Not completed — Participant convenience | 12 | 8
Period: Observational Period
Arm/Group | Rivaroxaban (Xarelto, BAY59-7939) | Enoxaparin/VKA
Started | 2206 (All participants who took any study medication and entered the observational period.) | 2197 (All participants who took any study medication and entered the observational period.)
Completed | 2165 | 2156
Not Completed | 41 | 41
Not completed — Protocol Violation | 0 | 2
Not completed — Withdrawal by Subject | 9 | 5
Not completed — Lost to Follow-up | 1 | 11
Not completed — Death | 27 | 20
Not completed — Study terminated by sponsor | 3 | 1
Not completed — Protocol driven decision point | 0 | 1
Not completed — Lack of Efficacy | 1 | 0
Not completed — Technical problems | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Rivaroxaban (Xarelto, BAY59-7939) | Enoxaparin/VKA | Total
Number analyzed (Participants) | 2419 | 2413 | 4832
Age, Continuous [Mean (Standard Deviation); unit: Years] — Intention-to-treat (ITT) population
  Years | 57.9 (17.3) | 57.5 (17.2) | 57.7 (17.3)
Age, Customized [Number; unit: Participants] — Intention-to-treat (ITT) population
  Participants
    18 - < 40 years | 410 | 432 | 842
    40 - < 60 years | 794 | 779 | 1573
    60 - < 75 years | 740 | 754 | 1494
    ≥ 75 years | 475 | 448 | 923
Sex: Female, Male [Count of Participants; unit: Participants] — Intention-to-treat (ITT) population
  Participants
    Female | 1309 | 1247 | 2556
    Male | 1110 | 1166 | 2276

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Symptomatic Recurrent Venous Thromboembolism [VTE] (i.e. the Composite of Recurrent Deep Vein Thrombosis [DVT] or Fatal or Non-fatal Pulmonary Embolism [PE]) Until the Intended End of Study Treatment
Description: All events were adjudicated and confirmed by a central independent adjudication committee blinded to treatment. Events were assessed based on either compression ultrasound (for DVT), venography (for DVT), spiral computed tomography (CT) scanning (for PE), pulmonary angiography (for PE), ventilation/perfusion lung scan (for PE), lung scintigraphy (for PE), autopsy (for fatal PE) or unexplained death for which DVT/PE could not be ruled out (for fatal PE), and/or case summaries.
Time Frame: 3-, 6-, or 12-month study treatment period
Population: The intention-to-treat (ITT) population consisted of all randomized participants with valid informed consent. Participants were analyzed according to the treatment assigned at randomization.
Measure: Number; unit: Percentage of participants
Arm/Group | Rivaroxaban (Xarelto, BAY59-7939) | Enoxaparin/VKA
Number analyzed (Participants) | 2419 | 2413
Percentage of participants | 2.1 | 1.8
Statistical Analysis 1: Comparison: Rivaroxaban (Xarelto, BAY59-7939) vs Enoxaparin/VKA; The rivaroxaban to comparator hazard ratio was computed with a 95% CI (confidence interval) (two-sided testing). Based on this model, rivaroxaban would be considered at least as effective as the comparator if the upper limit of the CI was less than 2.0; Test type: Non-Inferiority or Equivalence — Assuming equal efficacy, a total of 88 events will give a power of 90% to demonstrate that rivaroxaban is at least as effective as the comparator, considering a relative non-inferiority upper CI margin for the hazard ratio of 2.0 (two-sided alpha=0.05). The mean overall incidence for the primary efficacy outcome of 3% was expected and therefore 1465 patients per group would be needed. This number was to be adjusted based on the observed overall incidence of symptomatic recurrent VTE; p = 0.0026, Regression, Cox; Stratified by intend treatment duration, adjusted for presence of active malignancy at baseline; Hazard Ratio (HR) = 1.12, 95% CI 2-sided [0.75 to 1.68], Standard Error of Mean 0.2067 — The standard error of the log hazard ratio was estimated

2. Secondary Outcome: Percentage of Participants With the Composite Variable Comprising Recurrent DVT, Non-fatal PE and All Cause Mortality Until the Intended End of Study Treatment
Description: All events were adjudicated and confirmed by a central independent adjudication committee blinded to treatment. Events were assessed based on either compression ultrasound (for DVT), venography (for DVT), spiral computed tomography (CT) scanning (for PE), pulmonary angiography (for PE), ventilation/perfusion lung scan (for PE), lung scintigraphy (for PE), autopsy (for deaths), results/films/images of confirmatory testing, and/or case summaries.
Time Frame: 3-, 6-, or 12-month study treatment period
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Rivaroxaban (Xarelto, BAY59-7939) | Enoxaparin/VKA
Number analyzed (Participants) | 2419 | 2413
Percentage of participants | 4.0 | 3.4
Statistical Analysis 1: Comparison: Rivaroxaban (Xarelto, BAY59-7939) vs Enoxaparin/VKA; Stratified by intend treatment duration, adjusted for presence of active malignancy at baseline; Test type: Superiority or Other; p = 0.33, Regression, Cox — Nominal p-value; Hazard Ratio (HR) = 1.16, 95% CI 2-sided [0.86 to 1.56], Standard Error of Mean 0.1500 — The standard error of the log hazard ratio was estimated

3. Secondary Outcome: Percentage of Participants With an Event for Net Clinical Benefit 1 Until the Intended End of Study Treatment
Description: Net clinical benefit 1: composite of recurrent DVT or non-fatal or fatal PE, and major bleeding. Major bleeding was overt bleeding associated with 2 g/dL or greater fall in hemoglobin, leading to a transfusion of ≥2 units, occurring in a critical site or contributing to death. Net clinical benefit was considered greater in those participants with fewer composite events. All events were adjudicated and confirmed by a central independent adjudication committee blinded to treatment, based on either compression ultrasound, venography, spiral computed tomography scanning, pulmonary angiography, ventilation/perfusion lung scan, lung scintigraphy, autopsy or unexplained death for which DVT/PE could not be ruled out, results/films/images of confirmatory testing, and/or case summaries.
Time Frame: 3-, 6-, or 12-month study treatment period
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Rivaroxaban (Xarelto, BAY59-7939) | Enoxaparin/VKA
Number analyzed (Participants) | 2419 | 2413
Percentage of participants | 3.4 | 4.0
Statistical Analysis 1: Comparison: Rivaroxaban (Xarelto, BAY59-7939) vs Enoxaparin/VKA; Test type: Superiority or Other; p = 0.275, Regression, Cox — Nominal p-value; Stratified by intend treatment duration, adjusted for presence of active malignancy at baseline; Hazard Ratio (HR) = 0.85, 95% CI 2-sided [0.63 to 1.14], Standard Error of Mean 0.1499 — The standard error of the log hazard ratio was estimated

4. Secondary Outcome: Percentage of Participants With Recurrent PE Until the Intended End of Study Treatment
Description: All events were adjudicated and confirmed by a central independent adjudication committee blinded to treatment. Events were assessed based on spiral computed tomography scanning, pulmonary angiography, ventilation/perfusion lung scan, lung scintigraphy, autopsy or unexplained death for which DVT/PE could not be ruled out, results/films/images of confirmatory testing, and/or case summaries.
Time Frame: 3-, 6- or 12-month study treatment period
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Rivaroxaban (Xarelto, BAY59-7939) | Enoxaparin/VKA
Number analyzed (Participants) | 2419 | 2413
Percentage of participants | 1.4 | 1.2
Statistical Analysis 1: Comparison: Rivaroxaban (Xarelto, BAY59-7939) vs Enoxaparin/VKA; Test type: Superiority or Other; p = 0.55, Regression, Cox — nominal p-value; Stratified by intend treatment duration, adjusted for presence of active malignancy at baseline; Hazard Ratio (HR) = 1.16, 95% CI 2-sided [0.70 to 1.93], Standard Error of Mean 0.2570 — The standard error of the log hazard ratio was estimated

5. Secondary Outcome: Percentage of Participants With Recurrent DVT Until the Intended End of Study Treatment
Description: All events were adjudicated and confirmed by a central independent adjudication committee blinded to treatment. Events were assessed based on either compression ultrasound, venography, results/films/images of confirmatory testing, and/or case summaries.
Time Frame: 3-, 6- or 12-month study treatment period
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Rivaroxaban (Xarelto, BAY59-7939) | Enoxaparin/VKA
Number analyzed (Participants) | 2419 | 2413
Percentage of participants | 0.7 | 0.8
Statistical Analysis 1: Comparison: Rivaroxaban (Xarelto, BAY59-7939) vs Enoxaparin/VKA; Test type: Superiority or Other; p = 0.85, Regression, Cox — Nominal p-value; Stratified by intend treatment duration, adjusted for presence of active malignancy at baseline; Hazard Ratio (HR) = 0.94, 95% CI 2-sided [0.49 to 1.79], Standard Error of Mean 0.3289 — The standard error of the log hazard ratio was estimated

6. Secondary Outcome: Percentage of Participants With Clinically Relevant Bleeding, Treatment-emergent (Time Window: Until 2 Days After Last Dose)
Description: All events were adjudicated and confirmed by a central independent adjudication committee blinded to treatment. Clinically relevant bleeding included major bleeding (overt bleeding associated with 2 g/dL or greater fall in hemoglobin, leading to a transfusion of 2 or more units of packed red blood cells or whole blood, occurring in a critical site or contributing to death) and non-major bleeding associated with medical intervention, unscheduled physician contact, (temporary) cessation of study treatment, discomfort for the participants such as pain, or impairment of activities of daily life.
Time Frame: 3-, 6- or 12-month study treatment period
Population: The valid-for-safety analysis population consisted of all participants who were randomized with valid informed consent and received at least one dose of anticoagulant study treatment after randomization (i.e. enoxaparin, warfarin, acenocoumarol, rivaroxaban). Participants were analyzed according to the treatment they actually received.
Measure: Number; unit: Percentage of participants
Arm/Group | Rivaroxaban (Xarelto, BAY59-7939) | Enoxaparin/VKA
Number analyzed (Participants) | 2412 | 2405
Percentage of participants | 10.3 | 11.4
Statistical Analysis 1: Comparison: Rivaroxaban (Xarelto, BAY59-7939) vs Enoxaparin/VKA; Test type: Superiority or Other; p = 0.23, Regression, Cox — If the primary efficacy analysis shows that rivaroxaban is non-inferior to the comparator, the principal safety outcome was to be compared between treatment groups to maintain the overall type I error of 0.05 (2-sided) (a closed testing procedure); Stratified by intend treatment duration, adjusted for presence of active malignancy at baseline; Hazard Ratio (HR) = 0.90, 95% CI 2-sided [0.76 to 1.07], Standard Error of Mean 0.08756 — The standard error of the log hazard ratio was estimated

7. Secondary Outcome: Percentage of Participants With All Deaths
Description: All events were adjudicated and confirmed by a central independent adjudication committee blinded to treatment. Events were assessed based on either autopsy, results/films/images of confirmatory testing, and/or case summaries.
Time Frame: 3-, 6- or 12-month study treatment period
Population: as for outcome 6
Measure: Number; unit: Percentage of participants
Arm/Group | Rivaroxaban (Xarelto, BAY59-7939) | Enoxaparin/VKA
Number analyzed (Participants) | 2412 | 2405
Percentage of participants
  All post-randomization | 2.6 | 2.1
  Treatment-emergent (time window: 2 days) | 1.2 | 0.8
  Treatment-emergent (time window: 7 days) | 1.5 | 1.1

8. Secondary Outcome: Percentage of Participants With Other Vascular Events, On-treatment (Time Window: Until 1 Day After Last Dose)
Description: All pre-defined vascular events (ST segment elevation myocardial infarction, non ST segment elevation myocardial infarction, unstable angina, ischemic stroke, transient ischemic attack, non-central nervous system systemic embolism or vascular death) were adjudicated and confirmed by a central independent adjudication committee blinded to treatment. Events were assessed based results/films/images of confirmatory testing, and/or case summaries.
Time Frame: 3-, 6- or 12-month study treatment period
Population: as for outcome 6
Measure: Number; unit: Percentage of participants
Arm/Group | Rivaroxaban (Xarelto, BAY59-7939) | Enoxaparin/VKA
Number analyzed (Participants) | 2412 | 2405
Percentage of participants | 1.5 | 1.5

9. Other Pre Specified Outcome: Percentage of Participants With the Individual Components of Efficacy Outcomes Until the Intended End of Study Treatment
Description: All events were adjudicated and confirmed by a central independent adjudication committee blinded to treatment, based on either compression ultrasound, venography, spiral computed tomography scanning, pulmonary angiography, ventilation/perfusion lung scan, lung scintigraphy, autopsy or unexplained death for which DVT/PE could not be ruled out, results/films/images of confirmatory testing, and/or case summaries. Major bleeding was overt bleeding associated with 2 g/dL or greater fall in hemoglobin, leading to a transfusion of ≥2 units, occurring in a critical site or contributing to death.
Time Frame: 3-, 6- or 12-month study treatment period
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Rivaroxaban (Xarelto, BAY59-7939) | Enoxaparin/VKA
Number analyzed (Participants) | 2419 | 2413
Percentage of participants
  Death (PE) | 0.1 | 0.04
  Death (PE cannot be excluded) | 0.3 | 0.2
  Symptomatic PE and DVT | 0.0 | 0.1
  Symptomatic recurrent PE only | 1.0 | 0.8
  Symptomatic recurrent DVT only | 0.7 | 0.7
  Death (bleeding) | 0.2 | 0.2
  Death (cardiovascular) | 0.4 | 0.1
  Death (other) | 1.3 | 1.5
  Major bleeding | 1.4 | 2.4

10. Other Pre Specified Outcome: Percentage of Participants With Symptomatic Recurrent VTE (i.e. the Composite of Recurrent DVT or Fatal or Non-fatal PE) During Observational Period
Description: as for outcome 1
Time Frame: Up to 30 days after the last intake of study medication
Population: Participants entering the observational period were participants for whom the investigator indicated on the eCRF (electronic case report form) that the participant entered the observational period or had a confirmed event more than one day and up to 30 days after the last dose as a component of the respective composite outcome.
Measure: Number; unit: Percentage of participants
Arm/Group | Rivaroxaban (Xarelto, BAY59-7939) | Enoxaparin/VKA
Number analyzed (Participants) | 2211 | 2201
Percentage of participants | 0.9 | 0.7

11. Other Pre Specified Outcome: Percentage of Participants With the Composite Variable Comprising Recurrent DVT, Non-fatal PE and All Cause Mortality During Observational Period
Description: as for outcome 2
Time Frame: Up to 30 days after the last intake of study medication
Population: Participants entering the observational period were participants for whom the investigator indicated on the eCRF that the participant entered the observational period or had a confirmed event more than one day and up to 30 days after the last dose as a component of the respective composite outcome.
Measure: Number; unit: Percentage of participants
Arm/Group | Rivaroxaban (Xarelto, BAY59-7939) | Enoxaparin/VKA
Number analyzed (Participants) | 2213 | 2203
Percentage of participants | 2.1 | 1.5

12. Other Pre Specified Outcome: Percentage of Participants With an Event for Net Clinical Benefit 1 During Observational Period
Description: as for outcome 3
Time Frame: Up to 30 days after the last intake of study medication
Population: as for outcome 11
Measure: Number; unit: Percentage of participants
Arm/Group | Rivaroxaban (Xarelto, BAY59-7939) | Enoxaparin/VKA
Number analyzed (Participants) | 2212 | 2201
Percentage of participants | 1.2 | 1.2

13. Other Pre Specified Outcome: Percentage of Participants With Recurrent DVT During Observational Period
Description: as for outcome 5
Time Frame: Up to 30 days after the last intake of study medication
Population: as for outcome 11
Measure: Number; unit: Percentage of participants
Arm/Group | Rivaroxaban (Xarelto, BAY59-7939) | Enoxaparin/VKA
Number analyzed (Participants) | 2210 | 2201
Percentage of participants | 0.3 | 0.1

14. Other Pre Specified Outcome: Percentage of Participants With the Individual Components of Efficacy Outcomes During Observational Period
Description: as for outcome 9
Time Frame: Up to 30 days after the last intake of study medication
Population: as for outcome 11
Measure: Number; unit: Percentage of participants
Arm/Group | Rivaroxaban (Xarelto, BAY59-7939) | Enoxaparin/VKA
Number analyzed (Participants) | 2213 | 2203
Percentage of participants
  Death (PE) | 0.09 | 0
  Death (PE cannot be excluded) | 0 | 0.05
  Symptomatic PE and DVT | 0.09 | 0
  Symptomatic recurrent PE only | 0.5 | 0.5
  Symptomatic recurrent DVT only | 0.2 | 0.1
  Death (bleeding) | 0.09 | 0.09
  Death (cardiovascular) | 0.3 | 0.05
  Death (other) | 0.8 | 0.7
  Major bleeding | 0.3 | 0.5

15. Post Hoc Outcome: Percentage of Participants With an Event for Net Clinical Benefit 2 Until the Intended End of Study Treatment
Description: Net clinical benefit 2: composite of recurrent DVT or non-fatal or fatal PE, major bleeding (associated with 2 g/dL or greater fall in hemoglobin, leading to transfusion of ≥2 units, occurring in a critical site or contributing to death), cardiovascular death, myocardial infarction, stroke, and non CNS (central nervous system) systemic embolism. Net clinical benefit was considered greater in those participants with fewer composite events. All events were adjudicated and confirmed by a central independent adjudication committee blinded to treatment, based on either compression ultrasound (DVT), venography (DVT), spiral CT scanning (PE), pulmonary angiography (PE), ventilation/perfusion lung scan (PE), lung scintigraphy (PE), autopsy or unexplained death for which DVT/PE could not be ruled out, results/films/images of confirmatory testing, and/or case summaries.
Time Frame: 3-, 6- or 12-month study treatment period
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Rivaroxaban (Xarelto, BAY59-7939) | Enoxaparin/VKA
Number analyzed (Participants) | 2419 | 2413
Percentage of participants | 4.5 | 4.8

16. Post Hoc Outcome: Percentage of Participants With an Event for Net Clinical Benefit 2 During Observational Period
Description: as for outcome 15
Time Frame: Up to 30 days after the last intake of study medication
Population: as for outcome 11
Measure: Number; unit: Percentage of participants
Arm/Group | Rivaroxaban (Xarelto, BAY59-7939) | Enoxaparin/VKA
Number analyzed (Participants) | 2213 | 2201
Percentage of participants | 1.5 | 1.4

ADVERSE EVENTS:
Arm/Group | Rivaroxaban (Xarelto, BAY59-7939) | Enoxaparin/VKA
Serious Adverse Events (participants affected / at risk) | 504/2412 | 495/2405
Other Adverse Events (participants affected / at risk) | 1053/2412 | 1065/2405
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rivaroxaban (Xarelto, BAY59-7939) (N=2412) | Enoxaparin/VKA (N=2405)
Anaemia (Blood and lymphatic system disorders) | 14 | 6
Anaemia folate deficiency (Blood and lymphatic system disorders) | 1 | 0
Coagulopathy (Blood and lymphatic system disorders) | 0 | 2
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 | 0
Eosinophilia (Blood and lymphatic system disorders) | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1
Haemolytic anaemia (Blood and lymphatic system disorders) | 1 | 0
Hypercoagulation (Blood and lymphatic system disorders) | 1 | 0
Idiopathic thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 2
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1
Pernicious anaemia (Blood and lymphatic system disorders) | 1 | 0
Splenic haemorrhage (Blood and lymphatic system disorders) | 0 | 1
Splenic infarction (Blood and lymphatic system disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 0
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 1 | 2
Acute myocardial infarction (Cardiac disorders) | 6 | 10
Angina pectoris (Cardiac disorders) | 3 | 4
Angina unstable (Cardiac disorders) | 7 | 2
Arrhythmia (Cardiac disorders) | 2 | 1
Atrial fibrillation (Cardiac disorders) | 8 | 11
Atrial flutter (Cardiac disorders) | 1 | 1
Atrioventricular block (Cardiac disorders) | 0 | 1
Cardiac arrest (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 9 | 7
Cardiac failure acute (Cardiac disorders) | 4 | 2
Cardiac failure congestive (Cardiac disorders) | 4 | 5
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0
Cardiogenic shock (Cardiac disorders) | 1 | 0
Cardiomyopathy (Cardiac disorders) | 0 | 1
Cor pulmonale (Cardiac disorders) | 3 | 1
Cor pulmonale acute (Cardiac disorders) | 1 | 0
Cor pulmonale chronic (Cardiac disorders) | 1 | 1
Coronary artery disease (Cardiac disorders) | 1 | 8
Coronary artery stenosis (Cardiac disorders) | 0 | 1
Left ventricular failure (Cardiac disorders) | 1 | 0
Mitral valve incompetence (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1
Myocardial ischaemia (Cardiac disorders) | 0 | 2
Myocarditis (Cardiac disorders) | 0 | 1
Palpitations (Cardiac disorders) | 2 | 2
Pericardial effusion (Cardiac disorders) | 1 | 1
Pericardial haemorrhage (Cardiac disorders) | 1 | 2
Pericarditis (Cardiac disorders) | 2 | 0
Right ventricular failure (Cardiac disorders) | 3 | 0
Sick sinus syndrome (Cardiac disorders) | 0 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 2
Supraventricular tachycardia (Cardiac disorders) | 1 | 4
Tachycardia (Cardiac disorders) | 1 | 2
Ventricular fibrillation (Cardiac disorders) | 1 | 0
Ventricular tachycardia (Cardiac disorders) | 3 | 1
Coronary artery dissection (Cardiac disorders) | 0 | 1
Acute coronary syndrome (Cardiac disorders) | 0 | 1
Congestive cardiomyopathy (Cardiac disorders) | 2 | 0
Acute left ventricular failure (Cardiac disorders) | 1 | 0
Atrial septal defect (Congenital, familial and genetic disorders) | 1 | 0
Hydrocele (Congenital, familial and genetic disorders) | 1 | 0
Phimosis (Congenital, familial and genetic disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 3 | 4
Vertigo positional (Ear and labyrinth disorders) | 1 | 0
Deafness unilateral (Ear and labyrinth disorders) | 0 | 1
Sudden hearing loss (Ear and labyrinth disorders) | 1 | 1
Addison's disease (Endocrine disorders) | 1 | 0
Adrenal haemorrhage (Endocrine disorders) | 1 | 1
Diabetes insipidus (Endocrine disorders) | 0 | 1
Goitre (Endocrine disorders) | 0 | 2
Hyperparathyroidism primary (Endocrine disorders) | 0 | 1
Hyperthyroidism (Endocrine disorders) | 0 | 1
Amaurosis (Eye disorders) | 0 | 1
Cataract (Eye disorders) | 0 | 1
Diplopia (Eye disorders) | 1 | 0
Eye haemorrhage (Eye disorders) | 0 | 3
Eye pain (Eye disorders) | 0 | 1
Optic ischaemic neuropathy (Eye disorders) | 1 | 0
Retinal degeneration (Eye disorders) | 0 | 1
Retinal haemorrhage (Eye disorders) | 0 | 1
Vision blurred (Eye disorders) | 0 | 1
Age-related macular degeneration (Eye disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 4
Abdominal pain upper (Gastrointestinal disorders) | 1 | 4
Acute abdomen (Gastrointestinal disorders) | 0 | 1
Anorectal disorder (Gastrointestinal disorders) | 0 | 1
Ascites (Gastrointestinal disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 1 | 1
Colitis ischaemic (Gastrointestinal disorders) | 1 | 0
Colonic polyp (Gastrointestinal disorders) | 2 | 0
Colonic stenosis (Gastrointestinal disorders) | 1 | 0
Dental caries (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 1 | 0
Diverticulum (Gastrointestinal disorders) | 1 | 1
Diverticulum intestinal (Gastrointestinal disorders) | 1 | 0
Diverticulum oesophageal (Gastrointestinal disorders) | 1 | 0
Duodenal ulcer (Gastrointestinal disorders) | 2 | 0
Dyspepsia (Gastrointestinal disorders) | 2 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0
Gastric haemorrhage (Gastrointestinal disorders) | 0 | 1
Gastric perforation (Gastrointestinal disorders) | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 1 | 0
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 | 1
Gastritis (Gastrointestinal disorders) | 1 | 2
Gastritis haemorrhagic (Gastrointestinal disorders) | 1 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 7 | 5
Haematemesis (Gastrointestinal disorders) | 4 | 2
Haematochezia (Gastrointestinal disorders) | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 1 | 0
Hiatus hernia (Gastrointestinal disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 1 | 0
Intestinal fistula (Gastrointestinal disorders) | 1 | 0
Intestinal infarction (Gastrointestinal disorders) | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Large intestine perforation (Gastrointestinal disorders) | 1 | 2
Melaena (Gastrointestinal disorders) | 2 | 7
Nausea (Gastrointestinal disorders) | 2 | 0
Oesophageal ulcer (Gastrointestinal disorders) | 1 | 0
Oesophageal ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 6 | 6
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 1
Small intestinal perforation (Gastrointestinal disorders) | 0 | 1
Tooth loss (Gastrointestinal disorders) | 1 | 0
Umbilical hernia (Gastrointestinal disorders) | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 2
Vomiting (Gastrointestinal disorders) | 3 | 3
Intestinal polyp (Gastrointestinal disorders) | 0 | 1
Gastrointestinal dysplasia (Gastrointestinal disorders) | 1 | 0
Subileus (Gastrointestinal disorders) | 1 | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 3
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 | 2
Retroperitoneal haematoma (Gastrointestinal disorders) | 0 | 2
Intestinal haemorrhage (Gastrointestinal disorders) | 1 | 3
Abdominal hernia (Gastrointestinal disorders) | 1 | 0
Large intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Abdominal wall haematoma (Gastrointestinal disorders) | 0 | 2
Asthenia (General disorders) | 1 | 0
Chest discomfort (General disorders) | 1 | 0
Chest pain (General disorders) | 21 | 27
Cyst (General disorders) | 0 | 1
Death (General disorders) | 4 | 2
Fatigue (General disorders) | 2 | 0
Gait disturbance (General disorders) | 1 | 0
Granuloma (General disorders) | 0 | 1
Impaired healing (General disorders) | 0 | 1
Malaise (General disorders) | 1 | 0
Multi-organ failure (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 1 | 2
Pyrexia (General disorders) | 4 | 2
Sudden death (General disorders) | 3 | 1
General physical health deterioration (General disorders) | 3 | 2
Adverse drug reaction (General disorders) | 0 | 1
Drug intolerance (General disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 6 | 3
Implant site thrombosis (General disorders) | 0 | 1
Device deposit issue (General disorders) | 0 | 1
Bile duct stone (Hepatobiliary disorders) | 1 | 1
Biliary colic (Hepatobiliary disorders) | 1 | 0
Cholangitis (Hepatobiliary disorders) | 1 | 1
Cholecystitis (Hepatobiliary disorders) | 2 | 1
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 4 | 5
Hepatic failure (Hepatobiliary disorders) | 1 | 2
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 1
Hepatic pain (Hepatobiliary disorders) | 1 | 0
Hepatic steatosis (Hepatobiliary disorders) | 0 | 1
Hepatitis (Hepatobiliary disorders) | 0 | 1
Hepatitis acute (Hepatobiliary disorders) | 1 | 0
Hepatitis chronic active (Hepatobiliary disorders) | 1 | 0
Ischaemic hepatitis (Hepatobiliary disorders) | 1 | 0
Jaundice (Hepatobiliary disorders) | 1 | 0
Cytolytic hepatitis (Hepatobiliary disorders) | 1 | 0
Antiphospholipid syndrome (Immune system disorders) | 1 | 1
Drug hypersensitivity (Immune system disorders) | 0 | 1
Hypersensitivity (Immune system disorders) | 1 | 0
Sarcoidosis (Immune system disorders) | 1 | 0
Appendicitis (Infections and infestations) | 0 | 2
Bacteraemia (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 5 | 8
Bronchopneumonia (Infections and infestations) | 4 | 4
Bronchopulmonary aspergillosis (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 4 | 5
Cystitis (Infections and infestations) | 0 | 1
Diverticulitis (Infections and infestations) | 1 | 0
Endocarditis (Infections and infestations) | 1 | 0
Endocarditis bacterial (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 3 | 0
Gastroenteritis salmonella (Infections and infestations) | 1 | 0
Hepatitis A (Infections and infestations) | 0 | 1
Herpes simplex (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 0 | 2
Lobar pneumonia (Infections and infestations) | 4 | 1
Localised infection (Infections and infestations) | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 3 | 4
Lung abscess (Infections and infestations) | 0 | 1
Mastitis (Infections and infestations) | 1 | 0
Osteomyelitis (Infections and infestations) | 0 | 2
Pneumonia (Infections and infestations) | 22 | 21
Pneumonia mycoplasmal (Infections and infestations) | 0 | 1
Pneumonia primary atypical (Infections and infestations) | 0 | 1
Postoperative wound infection (Infections and infestations) | 0 | 1
Pyelonephritis (Infections and infestations) | 3 | 2
Pyelonephritis acute (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 13 | 2
Sinusitis (Infections and infestations) | 1 | 0
Skin infection (Infections and infestations) | 0 | 1
Tracheobronchitis (Infections and infestations) | 1 | 0
Tuberculosis (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 7 | 4
Viral rash (Infections and infestations) | 0 | 1
Wound infection (Infections and infestations) | 2 | 0
Urosepsis (Infections and infestations) | 2 | 2
Anal abscess (Infections and infestations) | 1 | 0
Neutropenic sepsis (Infections and infestations) | 1 | 0
Appendiceal abscess (Infections and infestations) | 0 | 1
Groin abscess (Infections and infestations) | 0 | 1
Abscess limb (Infections and infestations) | 0 | 1
Abscess soft tissue (Infections and infestations) | 1 | 0
Prostate infection (Infections and infestations) | 0 | 1
Skin bacterial infection (Infections and infestations) | 0 | 1
Abscess neck (Infections and infestations) | 0 | 1
Pneumonia necrotising (Infections and infestations) | 1 | 0
Subdiaphragmatic abscess (Infections and infestations) | 1 | 0
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 1 | 2
Biliary sepsis (Infections and infestations) | 0 | 1
Joint abscess (Infections and infestations) | 1 | 0
Wound infection staphylococcal (Infections and infestations) | 1 | 0
Intervertebral discitis (Infections and infestations) | 1 | 0
Lung infection (Infections and infestations) | 3 | 4
Respiratory tract infection (Infections and infestations) | 1 | 2
Cholecystitis infective (Infections and infestations) | 1 | 0
Device related infection (Infections and infestations) | 1 | 0
Infectious peritonitis (Infections and infestations) | 4 | 0
Alcohol poisoning (Injury, poisoning and procedural complications) | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 3 | 0
Cerebral haemorrhage traumatic (Injury, poisoning and procedural complications) | 1 | 0
Concussion (Injury, poisoning and procedural complications) | 1 | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 2 | 0
Fall (Injury, poisoning and procedural complications) | 4 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0
Fibula fracture (Injury, poisoning and procedural complications) | 1 | 1
Foot fracture (Injury, poisoning and procedural complications) | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 2
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 1
Kidney rupture (Injury, poisoning and procedural complications) | 0 | 1
Multiple injuries (Injury, poisoning and procedural complications) | 0 | 1
Operative haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 2 | 2
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1
Soft tissue injury (Injury, poisoning and procedural complications) | 0 | 2
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 0
Splenic haematoma (Injury, poisoning and procedural complications) | 0 | 1
Sternal fracture (Injury, poisoning and procedural complications) | 0 | 1
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 1 | 3
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 3
Subdural haemorrhage (Injury, poisoning and procedural complications) | 0 | 3
Tendon rupture (Injury, poisoning and procedural complications) | 1 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 0
Traumatic haematoma (Injury, poisoning and procedural complications) | 0 | 2
Anaemia postoperative (Injury, poisoning and procedural complications) | 0 | 1
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 0 | 1
Perirenal haematoma (Injury, poisoning and procedural complications) | 0 | 1
Traumatic fracture (Injury, poisoning and procedural complications) | 1 | 0
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 | 2
Contusion (Injury, poisoning and procedural complications) | 1 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 2 | 3
Incision site haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Brain contusion (Injury, poisoning and procedural complications) | 0 | 1
Cardiac valve replacement complication (Injury, poisoning and procedural complications) | 0 | 1
Postoperative ileus (Injury, poisoning and procedural complications) | 1 | 0
Procedural complication (Injury, poisoning and procedural complications) | 0 | 1
Joint injury (Injury, poisoning and procedural complications) | 2 | 0
Limb injury (Injury, poisoning and procedural complications) | 1 | 0
Chest injury (Injury, poisoning and procedural complications) | 0 | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 1
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 | 1
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 | 1
Activated partial thromboplastin time prolonged (Investigations) | 1 | 0
Alanine aminotransferase increased (Investigations) | 6 | 9
Aspartate aminotransferase increased (Investigations) | 1 | 1
Blood amylase increased (Investigations) | 1 | 0
Blood potassium increased (Investigations) | 1 | 0
C-reactive protein increased (Investigations) | 0 | 1
Coagulation time prolonged (Investigations) | 0 | 1
Coagulation time shortened (Investigations) | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 0 | 1
Haemoglobin decreased (Investigations) | 1 | 0
International normalised ratio abnormal (Investigations) | 0 | 1
International normalised ratio increased (Investigations) | 1 | 4
Liver function test abnormal (Investigations) | 4 | 9
Prostatic specific antigen increased (Investigations) | 1 | 1
Ultrasound liver abnormal (Investigations) | 1 | 0
Ejection fraction decreased (Investigations) | 0 | 1
Medical observation (Investigations) | 1 | 0
Transaminases increased (Investigations) | 2 | 2
Hepatic enzyme increased (Investigations) | 3 | 1
Acidosis (Metabolism and nutrition disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 2
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Failure to thrive (Metabolism and nutrition disorders) | 0 | 1
Gout (Metabolism and nutrition disorders) | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 2 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 2
Hypovolaemia (Metabolism and nutrition disorders) | 0 | 1
Shock hypoglycaemic (Metabolism and nutrition disorders) | 1 | 0
Metabolic disorder (Metabolism and nutrition disorders) | 0 | 1
Malnutrition (Metabolism and nutrition disorders) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 6
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 3
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 1 | 9
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 4 | 3
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 4 | 6
Osteolysis (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 | 1
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 2 | 0
Scoliosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 0 | 1
Temporomandibular joint syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1
Pseudarthrosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 3 | 1
Intervertebral disc compression (Musculoskeletal and connective tissue disorders) | 0 | 1
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 | 1
Spinal disorder (Musculoskeletal and connective tissue disorders) | 1 | 0
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 1 | 0
Acute lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Acute promyelocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Benign oesophageal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bile duct cancer non-resectable (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Breast cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 | 1
Fibroadenoma of breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Gallbladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0
Glioblastoma multiforme (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 4
Lung carcinoma cell type unspecified recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Lung squamous cell carcinoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant ascites (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Mesothelioma malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 4
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to pleura (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Multiple myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Myelofibrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Neoplasm prostate (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Ovarian germ cell teratoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Parathyroid tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Polycythaemia vera (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Prostate cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Prostatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 3
Small cell lung cancer stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
T-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 2
Histiocytosis haematophagic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Gastrointestinal stromal tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to peritoneum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Rectal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 4
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 7
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Colon neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Mantle cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Ovarian epithelial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Pelvic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Adrenal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Extranodal marginal zone B-cell lymphoma (MALT type) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Gastric neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Rectal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastatic gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Inflammatory pseudotumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Altered state of consciousness (Nervous system disorders) | 1 | 0
Amyotrophic lateral sclerosis (Nervous system disorders) | 1 | 1
Ataxia (Nervous system disorders) | 0 | 1
Carotid artery stenosis (Nervous system disorders) | 0 | 1
Cauda equina syndrome (Nervous system disorders) | 1 | 0
Cerebellar haemorrhage (Nervous system disorders) | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 4
Cerebral infarction (Nervous system disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Clumsiness (Nervous system disorders) | 1 | 0
Coma (Nervous system disorders) | 1 | 0
Convulsion (Nervous system disorders) | 2 | 3
Dementia Alzheimer's type (Nervous system disorders) | 0 | 1
Depressed level of consciousness (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 3 | 3
Encephalopathy (Nervous system disorders) | 0 | 1
Epilepsy (Nervous system disorders) | 2 | 1
Guillain-Barre syndrome (Nervous system disorders) | 1 | 0
Haemorrhage intracranial (Nervous system disorders) | 0 | 2
Headache (Nervous system disorders) | 3 | 4
Hepatic encephalopathy (Nervous system disorders) | 1 | 0
Leukoencephalopathy (Nervous system disorders) | 1 | 0
Loss of consciousness (Nervous system disorders) | 0 | 1
Migraine (Nervous system disorders) | 0 | 1
Nervous system disorder (Nervous system disorders) | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 2 | 0
Parkinsonism (Nervous system disorders) | 1 | 0
Presyncope (Nervous system disorders) | 0 | 1
Sciatica (Nervous system disorders) | 2 | 1
Spinal cord compression (Nervous system disorders) | 0 | 1
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 8 | 6
Tension headache (Nervous system disorders) | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 3 | 3
Balance disorder (Nervous system disorders) | 1 | 0
VIIth nerve paralysis (Nervous system disorders) | 0 | 1
Lacunar infarction (Nervous system disorders) | 0 | 1
Haemorrhagic transformation stroke (Nervous system disorders) | 1 | 0
Cerebrovascular insufficiency (Nervous system disorders) | 1 | 0
Radicular pain (Nervous system disorders) | 1 | 0
Ischaemic stroke (Nervous system disorders) | 13 | 5
Parkinson's disease (Nervous system disorders) | 1 | 0
Complex regional pain syndrome (Nervous system disorders) | 0 | 1
Post abortion haemorrhage (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 2
Alcohol abuse (Psychiatric disorders) | 0 | 1
Alcoholism (Psychiatric disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 5 | 3
Bipolar I disorder (Psychiatric disorders) | 1 | 1
Confusional state (Psychiatric disorders) | 0 | 1
Delusion (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 4 | 3
Mania (Psychiatric disorders) | 1 | 0
Panic attack (Psychiatric disorders) | 1 | 0
Suicide attempt (Psychiatric disorders) | 1 | 1
Mental status changes (Psychiatric disorders) | 0 | 1
Somatoform disorder (Psychiatric disorders) | 1 | 0
Mental disorder (Psychiatric disorders) | 0 | 1
Mental disorder due to a general medical condition (Psychiatric disorders) | 0 | 1
Acute prerenal failure (Renal and urinary disorders) | 1 | 0
Anuria (Renal and urinary disorders) | 0 | 1
Bladder dilatation (Renal and urinary disorders) | 0 | 1
Dysuria (Renal and urinary disorders) | 1 | 0
Glomerulonephritis membranous (Renal and urinary disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 8 | 11
Nephritis (Renal and urinary disorders) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 3
Nephropathy toxic (Renal and urinary disorders) | 0 | 1
Nephrotic syndrome (Renal and urinary disorders) | 1 | 0
Renal colic (Renal and urinary disorders) | 0 | 3
Renal cyst (Renal and urinary disorders) | 0 | 1
Renal failure acute (Renal and urinary disorders) | 2 | 4
Urinary retention (Renal and urinary disorders) | 2 | 0
Urinary tract disorder (Renal and urinary disorders) | 1 | 0
Urinary bladder polyp (Renal and urinary disorders) | 1 | 0
Renal mass (Renal and urinary disorders) | 0 | 1
Renal impairment (Renal and urinary disorders) | 1 | 1
Urethral stenosis (Renal and urinary disorders) | 0 | 2
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 1
Cervical dysplasia (Reproductive system and breast disorders) | 0 | 1
Cervical polyp (Reproductive system and breast disorders) | 0 | 1
Dysfunctional uterine bleeding (Reproductive system and breast disorders) | 1 | 0
Menorrhagia (Reproductive system and breast disorders) | 9 | 2
Metrorrhagia (Reproductive system and breast disorders) | 4 | 2
Ovarian cyst (Reproductive system and breast disorders) | 0 | 1
Priapism (Reproductive system and breast disorders) | 0 | 1
Prostatitis (Reproductive system and breast disorders) | 0 | 1
Uterine polyp (Reproductive system and breast disorders) | 0 | 1
Uterine prolapse (Reproductive system and breast disorders) | 1 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 4 | 0
Vulval disorder (Reproductive system and breast disorders) | 1 | 0
Genital haemorrhage (Reproductive system and breast disorders) | 1 | 0
Prostatic mass (Reproductive system and breast disorders) | 0 | 1
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 4
Asthma (Respiratory, thoracic and mediastinal disorders) | 4 | 2
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 9 | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 17 | 13
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 6 | 8
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Pharyngeal cyst (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 9 | 11
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 4
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 4 | 8
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 6 | 1
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Pulmonary infarction (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pulmonary venous thrombosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 | 5
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Mediastinal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Angioedema (Skin and subcutaneous tissue disorders) | 1 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1
Dermatitis exfoliative (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatomyositis (Skin and subcutaneous tissue disorders) | 1 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 1
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 0 | 1
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 | 1
Lichen planus (Skin and subcutaneous tissue disorders) | 1 | 0
Purpura (Skin and subcutaneous tissue disorders) | 1 | 0
Rash morbilliform (Skin and subcutaneous tissue disorders) | 1 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 1
Skin necrosis (Skin and subcutaneous tissue disorders) | 0 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 2 | 0
Miscarriage of partner (Social circumstances) | 1 | 0
Abortion induced (Surgical and medical procedures) | 2 | 3
Aortic aneurysm (Vascular disorders) | 1 | 2
Aortic aneurysm rupture (Vascular disorders) | 0 | 2
Aortic dissection (Vascular disorders) | 2 | 0
Aortic thrombosis (Vascular disorders) | 0 | 1
Circulatory collapse (Vascular disorders) | 1 | 0
Embolism arterial (Vascular disorders) | 0 | 1
Haematoma (Vascular disorders) | 4 | 4
Hypertension (Vascular disorders) | 1 | 3
Hypertensive crisis (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 3 | 1
Hypovolaemic shock (Vascular disorders) | 0 | 1
Iliac artery thrombosis (Vascular disorders) | 0 | 1
Orthostatic hypotension (Vascular disorders) | 1 | 0
Peripheral ischaemia (Vascular disorders) | 1 | 0
Temporal arteritis (Vascular disorders) | 0 | 1
Thrombophlebitis superficial (Vascular disorders) | 1 | 0
Vena cava thrombosis (Vascular disorders) | 1 | 0
Lymphocele (Vascular disorders) | 1 | 0
Intra-abdominal haematoma (Vascular disorders) | 0 | 1
Varicophlebitis (Vascular disorders) | 1 | 0
Arterial haemorrhage (Vascular disorders) | 0 | 1
Intra-abdominal haemorrhage (Vascular disorders) | 1 | 2
Paradoxical embolism (Vascular disorders) | 1 | 0
Distributive shock (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Rivaroxaban (Xarelto, BAY59-7939) (N=2412) | Enoxaparin/VKA (N=2405)
Constipation (Gastrointestinal disorders) | 146 | 141
Diarrhoea (Gastrointestinal disorders) | 128 | 132
Nausea (Gastrointestinal disorders) | 113 | 131
Chest pain (General disorders) | 179 | 181
Nasopharyngitis (Infections and infestations) | 188 | 195
Contusion (Injury, poisoning and procedural complications) | 95 | 133
Back pain (Musculoskeletal and connective tissue disorders) | 87 | 134
Pain in extremity (Musculoskeletal and connective tissue disorders) | 172 | 162
Headache (Nervous system disorders) | 196 | 177
Cough (Respiratory, thoracic and mediastinal disorders) | 160 | 179
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 156 | 147
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 229 | 205

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less